CLINICAL TRIAL: NCT04733001
Title: A Randomized, Open-label, Single Dose, 3-way Crossover Clinical Trial to Investigate the Effect of Food on the Pharmacokinetics of HSG4112 in Healthy Male Volunteers
Brief Title: A Study to Investigate the Effect of Food on the Pharmacokinetics of HSG4112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSG4112-P1-02
Record Dates: First submitted 2021-01-18; First posted 2021-02-01 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSG4112 Treatment Arm: Fasted (Experimental): Single oral dosing of HSG4112 480 mg under fasted conditions
  Interventions: Drug: HSG4112
- HSG4112 Treatment Arm: Low-Calorie Diet (Experimental): Single oral dosing of HSG4112 480 mg under low-calorie (400-500 kcal with 100-125 kcal fat) diet conditions
  Interventions: Drug: HSG4112
- HSG4112 Treatment Arm: High-Calorie Diet (Experimental): Single oral dosing of HSG4112 480 mg under high-calorie (800-1000 kcal with 500-600 kcal fat) diet conditions
  Interventions: Drug: HSG4112

INTERVENTIONS:
Drug: HSG4112 — Once-daily oral administration
  Other Names: 2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol

SUMMARY:
1. Study Objective: The objective of this clinical trial is to investigate the effect of food on the pharmacokinetics of HSG4112 after oral administration in healthy male subjects.
2. Study Design and Plan: This study is a randomized, open-label, single dose, 3-way crossover clinical trial. A unique randomization number will be assigned to each subject deemed eligible to participate in the study based on the inclusion/exclusion criteria. A total of 12 subjects will be randomized to 6 different sequence groups. Each subject will receive a single dose of HSG4112 480 mg via oral administration under fasted, low-fat diet, and high-fat diet conditions, with a washout period of 21 days in between each dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before screening.
2. Males between 19 and 50 years of age at screening.
3. Body mass index (BMI) between 18 and 26.9.

   ☞ BMI (kg/m2) = Body weight (kg) / {Height (m)^2}
4. In good health, determined by no clinically significant findings from medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory test at screening, or subjects who are deemed acceptable by the Investigator regardless of the test results.

Exclusion Criteria:

1. Significant history or clinical manifestation of any hepatic, kidney, neurological, immune, respiratory, endocrine, hematological, neoplastic, or cardiovascular disease, or psychiatric disorder (e.g., mood disorder, obsessive-compulsive disorder).
2. History of stomach or intestinal disorders (e.g., Chrons disease, ulcer) or surgeries - not including appendectomy, hemorrhoidectomy, or herniotomy - which may affect the safety or pharmacokinetic evaluation of the investigational product.
3. Significant history or clinical manifestation of hypersensitivity to any drug compound (e.g., licorice, aspirin, antibiotics).
4. One of more of the following laboratory test results at screening:

   * ALT (SGPT) > 60 IU/L
   * Glucose (fasting) > 110 mg/dL or < 70 mg/dL
   * Testosterone < 2.49 ng/mL or > 8.36 ng/mL
5. Systolic blood pressure of < 90 mmHg or > 150 mmHg, or diastolic blood pressure of < 60 mmHg or > 100 mmHg as determined by vital signs monitored after resting in sitting position for at least 3 minutes.
6. History of drug/chemical abuse or tested positive in urine drug screen.
7. Use or intend to use any prescription medications/products or phytotherapeutic/herbal/plant-derived preparations within 14 days prior to dosing, or any nonprescription medications/products (i.e., over-the-counter (OTC) drugs), health products, or vitamins within 7 days prior to dosing, unless deemed acceptable by the Investigator.
8. Participation in any clinical study or bioequivalence study involving administration of an investigational drug, including any study investigating HSG4112, within 6 months prior to dosing (i.e., within 6 months of the last dose from the previous study).
9. Whole blood donation within 2 months prior to dosing, plasma/platelet donation within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing.
10. Smoked > 10 cigarettes per day within 90 days prior to dosing.
11. Alcohol consumption of > 21 units/week (1 unit = 10 g of pure alcohol) or unable to abstain from consuming alcohol during the study period.
12. Ingestion of grapefruit-containing foods or beverages 24 hours prior to dosing until discharge, or unable to abstain from ingesting such foods or beverages during the same period.
13. Unable to abstain from caffeine-containing foods or beverages (e.g., coffee, tea (e.g., black tea, green tea), soft drinks, coffee milk, energy drinks, sports drinks) during the admission period.
14. Unable or unwilling to use acceptable contraceptive methods during the study period.

    ☞ Acceptable contraceptive methods include:
    * Use of an intrauterine device, which has been proven highly effective, by the subject's spouse/partner.
    * Physical contraception for subject or spouse/partner used with chemical sterilization.
    * Surgical sterilization (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy) of the subject or the subject's spouse/partner.
15. Subjects who, in the opinion of the Investigator, should not participate in this study based on clinical laboratory test results or other reasons.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval | Hour 0 to 24
  Area under the plasma concentration-time curve of HSG4112 over dosing interval (AUCtau)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point | Hour 0 to 192
  Area under the plasma concentration-time curve from time zero to the last measurable point (AUClast)
Pharmacokinetic Assessment by Maximum Plasma Concentration of HSG4112 | Hour 0 to 192
  Maximum plasma concentration of HSG4112 (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity | Hour 0 to 192
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf)
Pharmacokinetic Assessment by Time to Maximum Observed Plasma Concentration of HSG4112 | Hour 0 to 192
  Time to maximum observed plasma concentration of HSG4112 (Tmax)
Pharmacokinetic Assessment by Half-Life of HSG4112 | Hour 0 to 192
  Half-life of HSG4112 (T1/2)
Pharmacokinetic Assessment by Oral Clearance of HSG4112 | Hour 0 to 192
  Oral clearance of HSG4112 (CL/F)
Pharmacokinetic Assessment by Volume of Distribution of HSG4112 | Hour 0 to 192
  Volume of distribution of HSG4112 (Vd/F)

OTHER OUTCOMES:
Safety and Tolerability Assessment by Number of Participants with Change in Vital Signs | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in vital signs including blood pressure (mmHg) measured with blood pressure monitor, heart rate (beats per minute) measured with pulse oximeter, and body temperature (degrees Celcius) measured with thermometer
Safety and Tolerability Assessment by Number of Participants with Change in 12-Lead Electrocardiogram | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in 12-lead electrocardiogram
Safety and Tolerability Assessment by Number of Participants with Change in Laboratory Test | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in laboratory test assessed through hematology, blood biochemistry, urinalysis, and blood coagulation test
Safety and Tolerability Assessment by Number of Patients with Change in Physical Examination | Up to 3 weeks from day of last dosing
  Number of participants with clinically significant change in physical examination
Safety and Tolerability Assessment by Number of Patients with Change in Semen Volume | Up to 12 weeks from day of last dosing
  Pre-to-post examination of semen volume (milliliters) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Semen pH | Up to 12 weeks from day of last dosing
  Pre-to-post examination of semen pH by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Semen White Blood Cells | Up to 12 weeks from day of last dosing
  Pre-to-post examination of semen white blood cells (10^3 per microliter) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Sperm Count | Up to 12 weeks from day of last dosing
  Pre-to-post examination of sperm count (10^6 per milliliter) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Sperm Motility | Up to 12 weeks from day of last dosing
  Pre-to-post examination of sperm motility (percent of sperm with normal motility) by semen analysis to assess the safety and tolerability of HSG4112
Safety and Tolerability Assessment by Number of Patients with Change in Sperm Morphology | Up to 12 weeks from day of last dosing
  Pre-to-post examination of sperm morphology (percent of normal sperm) by semen analysis to assess the safety and tolerability of HSG4112

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No